CLINICAL TRIAL: NCT04471116
Title: Influence of OMNi-BiOTiC® FLORA Plus+ on the Vaginal Microbiome of Patients Suffering From Infertility
Brief Title: Influence of Probiotics on the Vaginal Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinderwunsch Institut GmbH (Other)
Collaborators: Institut AllergoSan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FRED002
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Vaginal Microbiome
Keywords: infertility; dysbiosis; probiotics; Lactobacillus; microbiome
MeSH Terms: conditions — Infertility; Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy group (Active Comparator): Patients in the therapy group took 1 sachet of OMNi-BiOTiC® FLORA plus + (= 2 g) dissolved in 1/8 l of water once a day
  Interventions: Dietary Supplement: OMNi-BiOTiC® FLORA plus+
- Control group (No Intervention): Patients in the control group received no additional medication.

INTERVENTIONS:
Dietary Supplement: OMNi-BiOTiC® FLORA plus+ — OMNi-BiOTiC® FLORA plus + is a dietary supplement for the treatment of a disturbed vaginal flora (dysbiosis). The product combines probiotic bacterial strains with a special fiber mixture. The product contains the following strains: Lactobacillus crispatus LBV88, Lactobacillus rhamnosus LBV96, Lactobacillus gasseri LBV150N and Lactobacillus jensenii LBV116
  Arms: Therapy group

SUMMARY:
The study aims to assess the influence of a probiotic supplement (OMNi-BiOTiC® FLORA plus +) on the vaginal microbiome composition of women suffering from infertility.

DETAILED DESCRIPTION:
Infertility is a global phenomenon affecting around 186 millions of people worldwide. Many circumstances have been identified to cause infertile conditions, with age being one of the most limiting factors. However, in recent years the microbiome has gained importance in the treatment of infertility and is considered as another important player to improve success rate of reproductive medicine treatments like in-vitro-fertilization (IVF).

Within the female reproductive tract the dominance of Lactobacilli is associated with a healthy vaginal microbial community in healthy reproductive-aged women. Since the microbiome has gained so much importance, its influence in IVF treatments is still controversially discussed. While some studies suggest a negative influence of vaginal dysbiosis on pregnancy rates a current meta-analysis showed no association between abnormal vaginal flora and conception rates following IVF treatment. One therapeutic approach is the administration of beneficial microorganisms (probiotics), mainly Lactobacillus species. The supplementation of exogenous lactobacilli strains has been suggested as cure for a dysbiotic vaginal flora to re-establish healthy conditions and improving female fertility health.

Hence, in the present study we wanted to investigate the impact of 4 probiotic strains (Lactobacillus crispatus LBV88, Lactobacillus rhamnosus LBV96, Lactobacillus gasseri LBV150N and Lactobacillus jensenii LBV116) on the relative abundance of vaginal microbiata species in women suffering from infertility.

80 infertile women suffering from infertility were included in the study within fertility treatment. 40 patients with IVF / ICSI were examined (20 with OMNi-BiOTiC® FLORA plus +, 20 as a control) and 40 patients with IUI / VZO (20 with OMNi-BiOTiC® FLORA plus +, 20 as a control). The control patients were selected from the routine patient collective of the Kinderwunsch Institut Schenk GmbH and receive no treatment with probiotics or placebo. Patients in the therapy group took 1 sachet of OMNi-BiOTiC® FLORA plus + (= 2 g) dissolved in 1/8 l of water once a day. Patients in the control group received no additional medication for routine treatment. Patients were randomized after inclusion in the study (block randomization).

On day 20 in the pre-cycle of hormonal stimulation, a vaginal smear sample was taken from the patient. The investigator introduced a sterile swab (eSwabTM, Copan Diagnostics Inc., USA), and took material from the mucosal surface. The eSwab was transferred to a sterile Falcon tube, stored at -72 ° C and then handed over to the company biovis Diagnostik MVZ GmbH (Germany) for 16s rRNA gene analysis. On day 20 in the stimulated cycle or subsequent cycle of the fertility treatment, another vaginal smear sample was taken and also stored in a sterile Falcon tube at -72 ° C.

The microbiota was determined using 16s rRNA gene analysis. The bacterial genomic DNA was isolated from the samples and the region V3-V4 was sequenced (Nextera XT, DNA Library Preparation Kit; Illumina MiSeq, Illumina, The Netherlands).

ELIGIBILITY:
Inclusion Criteria:

* patients with primary or secondary infertility
* age between 18 and 40
* signed informed consent
* BMI between 19 and 29.9

Exclusion Criteria:

* Patients with severe, acute and / or chronic diseases
* obesity
* hirsutism
* current intake of antibiotics
* State after hysterectomy
* Simultaneous use of other probiotics

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
vaginal microbiome | 1 month
  The microbiota was determined using 16s rRNA gene analysis. The bacterial genomic DNA was isolated from the samples and the region V3-V4 was sequenced

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schenk, MD, Principal Investigator — Kinderwunsch Institut GmbH
Locations (1):
- Das Kinderwunsch Institut Schenk GmbH, Dobl, Styria, Austria

IPD SHARING:
Plan to Share IPD: No
Data will be available within a publication of the study

REFERENCES:
- [Background] Inhorn MC, Patrizio P. Infertility around the globe: new thinking on gender, reproductive technologies and global movements in the 21st century. Hum Reprod Update. 2015 Jul-Aug;21(4):411-26. doi: 10.1093/humupd/dmv016. Epub 2015 Mar 22. PMID 25801630
- [Background] Moreno I, Codoner FM, Vilella F, Valbuena D, Martinez-Blanch JF, Jimenez-Almazan J, Alonso R, Alama P, Remohi J, Pellicer A, Ramon D, Simon C. Evidence that the endometrial microbiota has an effect on implantation success or failure. Am J Obstet Gynecol. 2016 Dec;215(6):684-703. doi: 10.1016/j.ajog.2016.09.075. Epub 2016 Oct 4. PMID 27717732
- [Background] Miles SM, Hardy BL, Merrell DS. Investigation of the microbiota of the reproductive tract in women undergoing a total hysterectomy and bilateral salpingo-oopherectomy. Fertil Steril. 2017 Mar;107(3):813-820.e1. doi: 10.1016/j.fertnstert.2016.11.028. Epub 2017 Jan 6. PMID 28069180
- [Background] Haahr T, Jensen JS, Thomsen L, Duus L, Rygaard K, Humaidan P. Abnormal vaginal microbiota may be associated with poor reproductive outcomes: a prospective study in IVF patients. Hum Reprod. 2016 Apr;31(4):795-803. doi: 10.1093/humrep/dew026. Epub 2016 Feb 23. PMID 26911864
- [Background] van Oostrum N, De Sutter P, Meys J, Verstraelen H. Risks associated with bacterial vaginosis in infertility patients: a systematic review and meta-analysis. Hum Reprod. 2013 Jul;28(7):1809-15. doi: 10.1093/humrep/det096. Epub 2013 Mar 29. PMID 23543384